CLINICAL TRIAL: NCT04560881
Title: Randomized, Double Blind, Placebo Parallel-controlled Phase III Clinical Trial to Evaluate the Efficacy, Immunogenicity and Safety of the Inactivated SARS-CoV-2 Vaccine (Vero Cell) in Argentine Healthy Population Aged Between 18 and 85 Years
Brief Title: Clinical Trial to Evaluate the Efficacy, Immunogenicity and Safety of the Inactivated SARS-CoV-2 Vaccine (COVID-19)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); China National Biotec Group Company Limited (Industry); Fundación Huésped (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BIBP2020003AR
Record Dates: First submitted 2020-09-16; First posted 2020-09-23 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: COVID-19 Virus Infection
Keywords: COVID-19; SARS-CoV-2 infection; Inactivated SARS-CoV-2 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 inactivated vaccines

STUDY DESIGN:
Intervention Model Description: Clinical trial conducted in randomized, double-blinded, placebo-controlled design.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inactivated SARS-CoV-2 vaccine, manufactured by BIBP (Experimental): Intramuscular injection
  Interventions: Biological: Inactivated SARS-CoV-2 vaccine (Vero cell)
- Placeboof Inactivated SARS-CoV-2 vaccine, manufactured by BIBP (Placebo Comparator): Intramuscular injection
  Interventions: Biological: Placebo/Aluminum Adjuvant of Inactivated SARS-CoV-2 vaccine

INTERVENTIONS:
Biological: Inactivated SARS-CoV-2 vaccine (Vero cell) — Immunization schedule: 2-doses of investigational vaccine or placebo are inoculated to the deltoid muscle of the upper arm according to the immunization schedule of Day 0, 21.
  Arms: Inactivated SARS-CoV-2 vaccine, manufactured by BIBP
Biological: Placebo/Aluminum Adjuvant of Inactivated SARS-CoV-2 vaccine — Immunization schedule: 2-doses of investigational vaccine or placebo are inoculated to the deltoid muscle of the upper arm according to the immunization schedule of Day 0, 21.
  Arms: Placeboof Inactivated SARS-CoV-2 vaccine, manufactured by BIBP

SUMMARY:
This is a randomized, double blind, placebo parallel-controlled phase III clinical trial to evaluate the efficacy, immunogenicity and safety of the inactivated SARS-CoV-2 Vaccine (Vero cell) in Argentine healthy population aged between 18 and 85 years old.

DETAILED DESCRIPTION:
SARS-CoV-2 belongs to β Coronavirus family and is a pathogen that can spread across races and is easy to cause respiratory diseases.

In December 2019, patients with pneumonia of unknown causes showed fever, cough, dyspnea, accompanied by medical imaging change of patchy diffuse infiltration of the lungs [2]. Through genome sequencing and analysis of lower respiratory tract alveolar lavage fluid samples from patients with pneumonia of unknown cause, a novel coronavirus different from any known virus was found. The World Health Organization WHO named the virus 2019 novel coronavirus, or 2019-nCoV for short, and the disease caused by the virus was named COVID-19. WHO listed the epidemic as a public health emergency of international concern.

With the spread of the SARS-CoV-2 epidemic in the world, vaccines have become the best weapon for epidemic prevention and control. At present, no vaccine to prevent coronavirus disease (COVID-19) in 2019 has been approved for listing. Based on the experience accumulated in the research and development of coronavirus vaccines in the past, the target of vaccines is also mainly focused on S protein.

Inactivated Virus Vaccine inactivates the virus obtained by culture by heating or chemical methods. The inactivated virus loses its pathogenicity and retains the main antigenic characteristics of the virus capsid, which can stimulate the specific immune response of human body. The inactivated SARS-CoV-2 vaccine (Vero cell) is prepared by inoculating African green monkey kidney cells (Vero cell) with the SARS-CoV-2 HB02 strain, culturing, harvesting, inactivating, clarifying, concentrating, purifying, and adding aluminum hydroxide adjuvant. After inoculating the vaccine, the recipients can produce immune response to prevent diseases caused by SARS-CoV-2. The inactivated SARS-CoV-2 vaccine (Vero cell) is prepared by inoculating African green monkey kidney cells (Vero cell) with the SARS-CoV-2 HB02 strain, culturing, harvesting, inactivating, clarifying, concentrating, purifying, and adding aluminum hydroxide adjuvant. After inoculating the vaccine, the recipients can produce immune response to prevent diseases caused by SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 18 and 85 years old.
* By asking for medical history and physical examination, the investigator judged that the health condition is well.
* Female subjects of childbearing age are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 3 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* During the whole follow-up period of the study, be able and willing to complete the whole prescribed study plan.
* With self-ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and be able to comply with the requirements of the protocol.

Exclusion Criteria:

* Active Sars-Cov-2 Infection measured by RT-qPCR
* Has a history of SARS, MERS infection (self-report, on-site inquiry)
* Has clinical manifestation of fever (axillary temperature > 37.0 ℃), dry cough, fatigue, nasal obstruction, runny nose, pharyngeal pain, myalgia, diarrhea, shortness of breath and dyspnea occurred within 14 days before vaccination.
* Body temperature > 37.0 ℃ before vaccination
* Urine pregnancy test positive;
* Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of inactivated SARS-CoV-2 vaccine have occurred.
* Has a history of convulsion, epilepsy, encephalopathy or mental illness or family history.
* With congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* With severe liver and kidney diseases, uncontrollable hypertension (systolic blood pressure ≥ 140 mmHg, diastolic blood pressure ≥ 90 mmHg), diabetic complications, malignant tumors, various acute diseases, or acute attack period of chronic diseases.
* Has been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, or other autoimmune diseases.
* With known or suspected diseases include severe respiratory diseases, severe cardiovascular diseases, liver and kidney diseases, and malignant tumors.
* Has a history of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease)
* Receiving anti-TB therapy.
* Patients receiving immunotherapy or inhibitor therapy within 3 months (continuous oral or infusion for more than 14 days)
* Inoculated live attenuated vaccines within 1 month before this vaccination, other vaccines are inoculated within 14 days before this vaccination.
* Received blood products within 3 months before this vaccination
* Received other research drugs within 6 months before this vaccination.
* Other circumstances judged by investigators that are not suitable for this clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Incidence of COVID-19 cases after two-doses of vaccination | 14 days after the full course of vaccination
  All confirmed COVID -19 cases 14 days after the full course of vaccination among healthy population aged between 18 and 85 years old.

SECONDARY OUTCOMES:
The 4-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 14 days after 2-dose of immunization and 28 days after full course of immunization
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 14 days after 2-dose of immunization and 28 days after full course of immunization
The Geometric Mean Increase (GMI) of anti-SARS-CoV-2 neutralizing antibody | 14 days after 2-dose of immunization and 28 days after full course of immunization
Incidence of any adverse reactions/events | Within 30 minutes after each dose of vaccine
Incidence of adverse reactions/events | 0 ~ 21/28 days after each dose of vaccine
Incidence of serious adverse events (SAE) | From the beginning of the first dose to 12 months after the whole course of immunization

OTHER OUTCOMES:
Anti-SARS-CoV-2 neutralizing antobody (NtAb) (immunological surrogate endpoint) | 14 days after 2-dose of immunization.
  The protective level of Anti-SARS-CoV-2 NtAbs

CONTACTS AND LOCATIONS:
Locations (4):
- Argentina (4):
  - Fundación Huésped, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Vacunar Liniers, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Vacunar Cañitas, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Vacunar Coghlan, Ciudad Autónoma de Buenos Aires, Buenos Aires